CLINICAL TRIAL: NCT01594814
Title: Patients' Perspective on Radiofrequency Catheter Ablation of AVRT and AVNRT - a Quality of Life, Utility and Willingness to Pay Study (PPRA Study)
Brief Title: Patients' Perspective on Radiofrequency Catheter Ablation of AVRT and AVNRT
Acronym: PPRA
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: PPRA
Record Dates: First submitted 2012-05-08; First posted 2012-05-09 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Tachycardia, Atrioventricular Nodal Reentry; Re-entrant Atrioventricular Tachycardia
Keywords: AVNRT; AVRT; WPW
MeSH Terms: conditions — Tachycardia, Atrioventricular Nodal Reentry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- RFA of AVNRT of AVRT
  Interventions: Procedure: RFA

INTERVENTIONS:
Procedure: RFA — radiofrequency ablation of slow pathway or accesory pathway

SUMMARY:
Atrioventricular nodal reciprocating tachycardia (AVNRT) and atrioventricular reciprocating tachycardia (AVRT) are two similar supraventricular re-entry tachycardias (SVT) emerging in relatively young age in patients without apparent structural heart disease or significant comorbidities. The treatment of choice in those patients is radiofrequency ablation (RFA).

The PPRA study is a prospective observational study developed to thoroughly analyze quality of life, utility and willingness-to-pay of Polish patients undergoing RF ablation of AVNRT or AVRT.

Based on collected data the investigators will prepare a profile of patient who will benefit most from radiofrequency ablation and who should be scheduled in first place for the ablation in case of problems with accessibility to this service.

What is more an analysis of medical and indirect costs of care will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age above 18
3. Scheduled RFA due to AVNRT or AVRT
4. Sufficient knowledge of the Polish language to independently complete the questionnaires

Exclusion Criteria:

1. No written informed consent
2. Health states significantly impairing QoL (eg. stroke, advanced heart failure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for ablation of AVNRT, AVRT or SVT will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2012-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (HRQOL) | two months
  Mean score of Patient Perception of Arrhythmia Questionnaire (PPAQ) - a disease-specific QoL questionnaire for patients suffering from supraventricular tachycardia translated and validated according to ISPOR (International Society For Pharmacoeconomics and Outcomes Research) guidelines

SECONDARY OUTCOMES:
Utility of health state | two months
  Mean score of EQ-5D - a generic questionnaire measuring a health state utility (official Polish translation)
Medical and indirect cost | one year
  Cross-sectional data gathered using original questionnaire designed to measure medical and indiresct costs related to arrhythmia incurred during a year preceding RFA
Willingness-to-pay | one day
  a cross-sectional willingness-to-pay questionnaire studying hypothetical situation where RFA was not financed by Polish Health Fund
Effectiveness | two days
  Data on medical history, final diagnosis, outcome of treatment, safety and future recommendations

CONTACTS AND LOCATIONS:
Overall Officials: Mariusz Pytkowski, MD, PhD, Study Chair — National Institute of Cardiology, Warsaw, Poland; Michal M Farkowski, MD, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- Institute of Cardiology, II Dept. of Coronary Heart Disease, Warsaw, Poland

REFERENCES:
- [Result] Farkowski MM, Pytkowski M, Maciag A, Golicki D, Wood KA, Kowalik I, Kuteszko R, Szwed H. Gender-related differences in outcomes and resource utilization in patients undergoing radiofrequency ablation of supraventricular tachycardia: results from Patients' Perspective on Radiofrequency Catheter Ablation of AVRT and AVNRT Study. Europace. 2014 Dec;16(12):1821-7. doi: 10.1093/europace/euu130. Epub 2014 Jun 11. PMID 24919538
- [Result] Farkowski MM, Pytkowski M, Golicki D, Szumowski L, Wood KA, Szwed H. Translation and cultural adaptation of a Patient Perception of Arrhythmia Questionnaire in Poland. Kardiol Pol. 2014;72(3):246-53. doi: 10.5603/KP.a2013.0318. Epub 2013 Dec 2. PMID 24293142
- [Derived] Farkowski MM, Pytkowski M, Maciag A, Golicki D, Kowalik I, Czech M, Rucinski P, Szwed H. Patient's age rather than severity of the arrhythmia influences the cost of medical treatment of atrioventricular nodal or atrioventricular reciprocating tachycardia. J Interv Card Electrophysiol. 2016 Nov;47(2):197-202. doi: 10.1007/s10840-016-0167-9. Epub 2016 Aug 3. PMID 27488509